CLINICAL TRIAL: NCT06104072
Title: Adding Computer-based Cognitive Training to Conventional Rehabilitation Can Affect Postural Stability , Locomotion and Cognition in Parkinson's Disease Patients
Brief Title: Effect of Adding Computerized Cognitive Training on Balance, Locomotion and Cognition in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Engy Badreldin Saleh Moustafa, PhD (Other)
Responsible Party: Sponsor-Investigator, Engy Badreldin Saleh Moustafa, PhD, Dr., Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004746
Record Dates: First submitted 2023-10-20; First posted 2023-10-27 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: Computer-Based Cognitive training; Parkinsonian Disease; Postural Stability; Gait
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Clinical trial, where the recruited patients will be randomly assigned into 2 equal groups ( GA & GB) using sealed envelopes. control group (GA) and study group (GB). Patients in (GA) will be treated by a designed physiotherapy program consisted of aerobic exercise on treadmill, stretching exercise, Proprioceptive neuromuscular facilitation (PNF) techniques, Graduated active exercises, gait training, Reciprocal and weight shifting exercises for 60 minutes/session. Patients in (GB) will be treated by computer-based cognitive training (30 minutes) in addition to the same physiotherapy program as GA (30 minutes).
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients participated will be masked about the type of intervention, where (GA) patients will receive PT program for 60 minutes, while patients in (GB) will receive computer -based REHACOM cognitive training (30 minutes) in addition to the same PT program as (GA)(30 minutes).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (GA) (Placebo Comparator): Patients in control group (GA) will be treated by a designed physiotherapy program consisted of aerobic exercise on treadmill, stretching exercise, Proprioceptive neuromuscular facilitation (PNF) techniques, Graduated active exercises, gait training, Reciprocal and weight shifting exercises for 60 minutes/session, 3 days/week for 8 consecutive weeks
  Interventions: Other: A Designed Physical Therapy Program
- Study group (GB) (Experimental): Patients in (GB) will be treated by computer-based cognitive training for 30 minutes followed by the same physiotherapy program as GA for another 30 minutes. so the whole duration of the treatment session for (GB) is 60 minutes ( half of the session the computerized cognitive training and the other half is for the designed physical therapy program). the whole treatment intervention will be 3 days /week for 8 consecutive weeks.
  Interventions: Device: REHACOM Software; Other: A Designed Physical Therapy Program

INTERVENTIONS:
Device: REHACOM Software — It is a computer-based cognitive rehabilitation test that includes 32 cognition training tasks for attention/concentration, reaction behavior, memory , logical reasoning & executive functioning with graded difficulty . It is composed of regular PC , 1G RAM , DVD drive, 100 GB hard drive with windows XP SP3, 128 MB RAM direct 3D graphic card , Screen at least 19" , regular PC keyboard or Rehacom panel & printer .The Rehacom software version is (patientenpult (1990-1997) EN/ISO-13485-certified).
  * For each Cognitive training domain there is one hundred levels of difficulty.
  * Each patient is evaluated from level one(1) ang gradually increase the difficulty till we reach the level that will be used in the treatment sessions as the patient's performance improve we can proceed to the next level.
  * The period of the session was chosen to be maximum (60 minutes) for each patient with five minutes rest in between each level.
  Other Names: Computer-Based Cognitive Training
  Arms: Study group (GB)
Other: A Designed Physical Therapy Program — A designed physiotherapy program consisted of aerobic exercise on treadmill, stretching exercise, Proprioceptive neuromuscular facilitation (PNF) techniques, Graduated active exercises, postural correction, gait training, balance training on different base of supports using static and dynamic balance training with reciprocal and weight shifting exercises.

SUMMARY:
BACKGROUND: Postural instability and gait abnormalities are cardinal features in Parkinson's disease (PD). It represents one of the most disabling symptoms in the advanced stages of the disease.

The purpose of this study was to evaluate the immediate and long-term effects of adding computer-based cognitive training to physical therapy interventions on postural stability, locomotion, and cognitive performance in Parkinson's disease patients.

DETAILED DESCRIPTION:
Study design: A randomized control clinical trial among sixty-eight Egyptian Parkinson's Disease patients of both sexes participated in the study; their ages ranged from 55 to 70 years. They were selected from the Neurology Clinics and from the Movement Disorder Clinic, Neurology Department, Faculty of Medicine, Cairo University, in the period from May 2024 to March 2025.

The patients will be divided into two equal groups: the control group (GA) and the study group (GB). Patients in GA will be treated by a designed physiotherapy program consisting of aerobic exercise on a treadmill, stretching exercises, proprioceptive neuromuscular facilitation (PNF) techniques, graduated active exercises, gait training, reciprocal, and weight-shifting exercises for 60 minutes. Patients in (GB) will be treated with computer-based cognitive training using REHACOM (30 minutes) in addition to the same physiotherapy program as GA (30 minutes). Rehacom software will be used for cognitive training targeting four main cognitive domains; attention/concentration, figural memory, auditory response control, and visual response control. . The treatment session for all patients in both groups will be 60minutes/session. The whole treatment protocol will include 24 sessions, three sessions per week, for two successive months.

Primary Outcomes:

1. Postural stability:

   - Biodex balance system was used to assess dynamic balance indices ( Overall stability index, mediolateral stability & anteroposterior stability)
2. Spatio-temporal gait parameters:

   * Digital video camera and kinovea (video motion analysis software) was used to assess spatiotemporal gait parameters (Stride length, velocity & Cadence).

Secondary Outcome:

a. Overall cognitive functions:

- Parkinson's Disease - Cognitive Rating Scale (PD-CRS).

ELIGIBILITY:
Inclusion Criteria:

* Egyptian Parkinson's Disease patients of both sex , all patients fulfilled the U.K Parkinson's Disease Brain Bank Criteria for diagnosis of idiopathic PD.
* The patients' age ranged from 58 to 68 years.
* The duration of illness ranged from two to five years.
* The severity of the disease ranged from mild to moderate disability according to UPDRS motor scores (part III) and Modified Hoehn and Yahr staging (stage 2.5&3) .
* Cognitive function ranged from 65 to 81 according to Parkinson's Disease-Cognitive Rating Scale (PD-CRS) that indicates mild cognitive impairment.
* The patients with mild balance and gait impairments
* Medically and psychologically stable patients and of adequate cardiac function to adhere to the protocol.

Exclusion Criteria:

* Patients with secondary parkinsonism (Drug-induced, post traumatic, or post infectious) or atypical parkinsonism.
* Patients with major language disturbance, severe physical, auditory or visual impairment affecting their ability to complete testing.
* Patients with magnetic devices or any other implanted device (e.g., metallic implants such as pacemakers, surgical aneurysm clips…etc).
* Patients with a history of seizure, head injury or brain surgery.
* Complicating or unstable cardiovascular disease (unstable angina, recent myocardial infarction within the last three months, congestive heart failure, significant heart valve dysfunction, or unstable hypertension) or pulmonary disorders.
* Patients with musculoskeletal disorders such as severe arthritis, knee surgery, total hip joint replacement, lower limb fractures or contractures of fixed deformity.
* Patients with evidence from the history, physical examination, or special investigations for any concomitant medical or metabolic illness known to affect cognition e.g. cerebrovascular stroke, thyroid or parathyroid disease, hepatic or renal failure.
* Patients receiving certain drugs known to improve cognition (e.g. rivastigmine, memantine…..etc).
* Patients with current or prior history of major psychiatric disorder and/or current use of anxiolytic, neuroleptic, sedative medication or sleeping aids.
* Uncooperative patients.
* Illiterate patients.

Ages: 58 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-04-20 (Estimated)

PRIMARY OUTCOMES:
Overall Stability Index | Baseline Assessment, Immediately Post Treatment, 3 Month Posttreatment Assessment (Follow-up)
  o Overall balance index: represents the patient's ability to control balance in all directions. High values indicate balance disturbance (increase rate of body swaying during the test).
Anterior / posterior (A/P) index | Baseline Assessment, Immediately Post Treatment, 3 Month Posttreatment Assessment (Follow-up)
  o Anterior / posterior (A/P) index represents the patient's ability to control balance in front to back direction.
Medial/ lateral (M/L) index | Baseline Assessment, Immediately Post Treatment, 3 Month Posttreatment Assessment (Follow-up)
  o Medial/ lateral (M/L) index: represents the patient's ability to maintain balance from side to side.
Velocity of Gait | Baseline Assessment, Immediately Post Treatment, 3 Month Posttreatment Assessment (Follow-up)
  Using 2D motion analysis in Kinovea program for spatiotemporal gait analysis
  o Velocity = Distance/Time
  * The total distance: represented by the actual length that the patient walked and this was presented by the blue line (three meters).
  * The total duration of walking (seconds): was calculated by using the ''stop watch'' tool in kinovea program. Velocity meter/seconds: was calculated by dividing the total distance that had been walked by the patient over the total duration.
Cadence of Gait | Baseline Assessment, Immediately Post Treatment, 3 Month Posttreatment Assessment (Follow-up)
  Using 2D motion analysis in Kinovea program for spatiotemporal gait analysis Cadence is the Number of steps/Minute
  * Number of steps: calculated by counting the steps the patient walked from the beginning to the end of the walkway (blue line).
  * Cadence was calculated by dividing the number of steps that the patient walked over the actual duration of walking.
Stride Length | Baseline Assessment, Immediately Post Treatment, 3 Month Posttreatment Assessment (Follow-up)
  Using 2D motion analysis in Kinovea program, stride length was the distance from the first initial contact of one foot (1st frame) to the next initial contact of the ipsilateral foot (2nd frame).

SECONDARY OUTCOMES:
Overall cognitive performance | Baseline Assessment, Immediately Post Treatment, 3 Month Posttreatment Assessment (Follow-up)
  * Parkinson's Disease - Cognitive Rating Scale (PD-CRS) was conducted for each patient from a comfortable sitting position on a chair with back support and suitable seat height compared to a table in front of the patient.
  * The following cognitive domains were assessed: - Immediate free recall verbal memory (12 points), Confrontation naming (20 points), - Sustained attention (ten points), Working memory (ten points), - Visuo-constructional skills (Unprompted drawing of a clock) (ten points), Visuo-perceptual skills (Copy drawing of a clock) (ten points), - Delayed free recall verbal memory (12 points),Alternating verbal fluency (20 points) and - Action verbal fluency (30 points).
  The overall total score for the (PD-CRS) is 134, the lower the score the more the cognitive impairment. The inclusion criteria for PD patients with cognitive decline indicated that a score 65-84 was the optimal cutoff point on the total score for the PD-CRS indicating mild cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Engy B Saleh, PhD, Principal Investigator — Faculty of Physical Therapy, Cairo University, Egypt
Locations (1):
- Faculty of Physical Therapy, Cairo University, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No